CLINICAL TRIAL: NCT07344909
Title: The Effects of Essix Splint Therapy on Burning Mouth Syndrome. A Prospective N-of-1 Study.
Brief Title: Burning Mouth Syndrome: Effects of Occlusal Splint Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-04647-02
Record Dates: First submitted 2025-11-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Burning Mouth Syndrome; Orofacial Pain; Mouth Dryness
MeSH Terms: conditions — Burning Mouth Syndrome; Facial Pain; Xerostomia

STUDY DESIGN:
Intervention Model Description: N-of-1 design. Two two-week treatment arms with a one-week wash-out period in between.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essix splint (Experimental): The treatment (intraorally applied Essix splint) effect on pain and saliva. Each participant will use the Essix appliance and collect saliva together with a clinical examination and saliva collection at the clinic. A questionary will also be completed.
  Interventions: Device: Essix splint
- No Essix splint (No Intervention): Effect on pain and saliva while not using the splint: collection of saliva together with a clinical examination and saliva collection at the clinic. A questionary will also be completed.

INTERVENTIONS:
Device: Essix splint — The treatment effect of an intraorally applied Essix splint compared with periods without splint use. Each participant will use the Essix appliance and have a no-appliance period in randomized order
  Arms: Essix splint

SUMMARY:
Burning Mouth Syndrome (BMS) causes chronic oral pain and significantly affects quality of life. Effective treatments are limited and often provide only temporary relief.

This prospective N-of-1 study evaluates the effect of an intraoral Essix appliance on pain intensity and salivary secretion in patients with BMS.

Saliva samples are collected and analysed for volume and composition.

DETAILED DESCRIPTION:
Burning Mouth Syndrome often causes substantial suffering, both due to persistent oral pain and its long-term impact on quality of life, daily activities, and psychological well-being (including depression, anxiety, and stress). Effective treatment options for BMS remain limited, and existing interventions generally demonstrate only modest and temporary benefits.

This study aims to investigate the effect of an Essix appliance on pain relief and salivary secretion in patients with Burning Mouth Syndrome (BMS) using an N-of-1 design, in which each participant serves as their own control.

This is a prospective N-of-1 study designed to assess the treatment effect of an intraorally applied Essix splint compared with periods without splint use. Each participant will use the Essix appliance and have a no-appliance period in randomized order, each lasting one week, separated by a one-week washout period. During the active weeks, saliva samples (both unstimulated and chewing-stimulated) will be collected at home. Additionally, saliva will be collected twice at the Faculty of Odontology in randomized order.

Saliva samples will be analyzed for total protein concentration, with specific focus on lubricating glycoproteins (mucins) using antibody-based methods. Further analyses will employ lectins recognizing specific carbohydrate structures to characterize the glycosylation patterns of salivary glycoproteins and salivary markers.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral mucosal pain from participants in the previous BMS validation study.
* greater than 30% pain relief during prior use of an Essix appliance.
* chronic intraoral pain lasting more than 3 months.
* age between 18 and 80 years.

Exclusion Criteria:

* fibromyalgia
* ongoing dental treatment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Subjective change in pain perception | two weeks for wearing the splint and two weeks not wearing the splint. The time point for the measurement is during the two clinical appointments - directly after the period with the splint and directly after the period without the splint.
  Subjective perception of the change of pain in percent when wearing the splint and not wearing the splint
Saliva volume | Twice during the clinical appointments:one directly after the period of 2 weeks after using the splint and the another period directly after 2 weeks when not using the splint; and 8 times collection at home. Saliva collection in the morning hours.
  Saliva volume (rest saliva and stimulated saliva) in milliliters; 10 minutes collection for the rest saliva and 5 minutes collection for the stimulated saliva.
Concentration of glycoproteins in rest saliva | Two occasions -directly after the period of using the splint and after the period of not using the splint. The saliva is collected and then put into the freezer immediately. Analysis starts when whole saliva collection of all participants is finished.
  Glycoproteins from the rest saliva measured in mg/mL
Concentration of proteins in stimulated saliva | Stimulated saliva is collected in two occasions - periods with and without the splint. After the collection saliva is centrifuged immediately and then put into the freezer. Analysis starts when the whole collection is done.
  Saliva proteins e.g., inflammation-, stress-, or metabolism-related biomarkers from the stimulated saliva, measured in ng/mL.

SECONDARY OUTCOMES:
Global impression of change | Twice: after the time period with the splint (two weeks) and after the time period without the splint (two weeks). The score is taken during the clinical appointments - directly after the period with and without the splint.
  Subjective change of the condition using Patient Global Impression of Change Scale which scores the global perception of change: the scale is composed of expressions for change, starting with "Very much improved" and ending with "Very much worsened". The first one indicate a positive change and the later indicates a negativ change.
Subjective perception of mouth dryness | The score is taken twice: immediatle after the period with the splint (two weeks) and after the period without the splint (two weeks) - during the clinical appointments.
  Subjective description of the perceived mouth dryness using a numeric scale 0-10 where 0 indicates very dry and 10 indicates no dryness.

CONTACTS AND LOCATIONS:
Locations (1):
- Malmö university, Malmo, Sweden